CLINICAL TRIAL: NCT00733421
Title: The Effect of Anti-inflammatory Analgesics on Bone Repair, Pain and Gastro-intestinal Side Effects After Hallux Valgus Surgery; a Prospective Randomised Double-blind Placebo Controlled Study.
Brief Title: The Effect of Anti-inflammatory Analgesics on Pain Following Hallux Valgus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Jan Jakobsson, Foot & Ancle Surgical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008HV001; EudraCT number 2008-000791-24
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Results first posted 2010-01-13 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-08

CONDITIONS: Postoperative Pain
Keywords: Day surgery; Hallux Valgus; Pain; Analgesics
MeSH Terms: conditions — Pain, Postoperative; Hallux Valgus; Pain | interventions — Etoricoxib; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Active study drug:
  Etoricoxib 90 mg once daily
  Interventions: Drug: etoricoxib
- 2 (Active Comparator): Tramadol 100 mg slow release twice daily
  Interventions: Drug: tramadol

INTERVENTIONS:
Drug: etoricoxib — 90 mg once daily
  Other Names: Arcoxia
  Arms: 1
Drug: tramadol — 100 mg twice daily
  Other Names: Tiparol
  Arms: 2

SUMMARY:
The effects of none-steroidal anti-inflammatory drugs (NSAIDs) and selective cyclooxygenase inhibitors (Coxibs) on the formation of bone and fracture healing have been a matter of debate since long.

There is, however, limited data in humans and further prospective randomised studies are warranted. Ekman et al studied in a prospective randomised double blind study the effects of celecoxib, a selective cox-II-inhibitor, on pain and bone healing following spine surgery. They found significant effects on reduction of pain and need for opioid analgesics postoperatively but could see no negative effects the numbers of "none-unions" at a 1-year follow up 3.

In a similar prospective randomised double-blind study design significant effects in reduction of pain and need for rescue analgesia was seen from the use of celecoxib in the perioperative multi-modal pain strategy for cruciate-ligament reconstruction and no negative effects could bee seen on six month follow-up of the strength of the reconstructed ligament.

The aim of the present study is to further study the effects of the perioperative use of etoricoxib, a selective cox-II-inhibitor (Coxibs), in a prospective randomised double-blind study on bone healing, pain and need for rescue analgesia in patients undergoing elective Hallux Valgus surgery with a standardised surgical technique including an osteotomy of metatarsale I and excision of exostosis.

Study population 100 American Society of Anesthesiology (ASA) physiological status1-2 patients scheduled for elective hallux valgus (HV) surgery

The patients are going to be randomised into 2 groups, 50 patients in each;

1. etoricoxib 90 mg once daily x 5
2. tramadol 100 mg twice daily x 5

First line rescue medication t. paracetamol 1 gr up to 4 gram daily Second line rescue t. oxycodone 10 mg

Primary study variables:

* X-ray evaluation (computer tomography (CT)-investigation) of bone healing assessed a CT-scan modelling of the osteotomy at twelve weeks after surgery
* Number of patients requiring rescue medication
* Patient assessment using "brief pain inventory" 24 hours and 2 weeks after surgery

Secondary study variables are;

* Visual Analogue Scale (VAS) grading Day 1-7
* Compliance to base medication
* Need for rescue analgesia Day 1-7
* Adverse Effects

  * Experience of any emetic symptoms
  * Experience of any gastrointestinal symptoms
* Satisfaction with pain medication Day 20
* Wound dressing Day 20
* Clinical evaluation 17 weeks, final assessment

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* Health ASA 1-2 patients 18-65 years of age

Exclusion Criteria:

* ASA/NSAID allergy
* Renal disease
* Lithium therapy
* Complicated cardiovascular disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jakobsson, MD, PhD,, Principal Investigator — Foot & Ancle Surgical Center
Locations (1):
- Foot & Ancle Surgical Center, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patient recruited and analysed between october 2008 and june 2009
Pre-assignment Details: Two patients were excluded after randomization forgot study medication and questionnaire leaving the hospital
Groups:
- Etoricoxib: Active study drug:
  Etoricoxib 90 mg once daily
- Control Tramadol: Tramadol 100 mg slow release twice daily
Period: Overall Study
Arm/Group | Etoricoxib | Control Tramadol
Started | 50 (November 2008) | 50 (November 2008)
Completed | 49 (All but one randomsied patient) | 49 (All but one randomised patient)
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etoricoxib | Control Tramadol | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Requiring Rescue Medication
Description: Number of patients requiring any further pain medication
Time Frame: 7 day study period
Measure: Number; unit: patients
Arm/Group | Etoricoxib | Control Tramadol
Number analyzed (Participants) | 49 | 49
patients | 29 | 36

2. Secondary Outcome: Summary of Pain Scores, Day 1-7 of Visual Analogue Scale Grading of Pain
Description: VAS score 1-10 1=no pain 10 = worst possible pain, summary variable day 1-7; 7 - 70
Time Frame: The first 7 days after surgery, during study pain medication
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Etoricoxib | Control Tramadol
Number analyzed (Participants) | 49 | 49
scores on a scale | 12 (8) | 17 (11)

3. Secondary Outcome: Compliance to Base Medication
Description: Number of patients that did not discontinue study medication before day 7
Time Frame: 7-day study period, during study medication
Measure: Number; unit: patients
Arm/Group | Etoricoxib | Control Tramadol
Number analyzed (Participants) | 49 | 49
patients | 49 | 43

4. Secondary Outcome: Gastro-intestinal Symptoms
Description: Number of patients reporting any gastro-intestinal side effects; nausea and or vomiting, gastritis etc. assessed by patient and documented in written questionnaire
Time Frame: during the 7- day pain medication period
Measure: Number; unit: patients
Arm/Group | Etoricoxib | Control Tramadol
Number analyzed (Participants) | 49 | 49
patients | 6 | 20

5. Secondary Outcome: Dizziness/Sleepiness
Description: Number of patients that experienced dizziness/sleepiness/fatigue, assessed by patient and documented in written questionnaire
Time Frame: During the 7-day pain medication period
Measure: Number; unit: patients
Arm/Group | Etoricoxib | Control Tramadol
Number analyzed (Participants) | 49 | 49
patients | 2 | 13

6. Secondary Outcome: Wound Healing
Description: healing process assessed by a blinded physician during the final outpatient clinic visit assessment graded; Good/neutral/bad
Time Frame: 16 week follow-up
Measure: Number; unit: patients
Arm/Group | Etoricoxib | Control Tramadol
Number analyzed (Participants) | 42 | 47
patients
  Goood | 37 | 39
  Neutral | 5 | 6
  Bad | 0 | 2

7. Secondary Outcome: Satisfaction With Pain Medication
Description: satisfied or unsatisfied with study medication, assessed by patient in questionnaire
Time Frame: during the first 20 days after surgery, 1st outpatient clinic visit
Measure: Number; unit: patients
Arm/Group | Etoricoxib | Control Tramadol
Number analyzed (Participants) | 49 | 49
patients
  Satisfied | 47 | 39
  Not satisfied | 2 | 10

8. Secondary Outcome: Patient Assessed Overall Satisfaction With Surgery/Outcome
Description: overall satisfaction with outcome, patients assessed satisfaction with the surgical procedure; satisfied, neutral or unsatisfied, written questionnaire.
Time Frame: 16 weeks
Measure: Number; unit: Patients.
Arm/Group | Etoricoxib | Control Tramadol
Number analyzed (Participants) | 49 | 49
Patients.
  satisfied | 45 | 44
  neutral | 4 | 4
  unsatisfied | 0 | 1

9. Secondary Outcome: Patient Assessed Quality of Life
Description: Quality of Life evaluated by grading on a Visual Analogue Scale in the written questionnaireisual analogue scale grading 0-100; 0 death and 100 perfect quality of life
Time Frame: At 16-week post surgery follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Etoricoxib | Control Tramadol
Number analyzed (Participants) | 48 | 49
score on a scale | 94.5 (9.4) | 94.7 (7.8)

ADVERSE EVENTS:
Arm/Group | Etoricoxib | Control Tramadol
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 8/49 | 35/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoricoxib (N=49) | Control Tramadol (N=49)
Nausea (Gastrointestinal disorders) | 6 (6) | 20 (20)
dizziness (Nervous system disorders) | 2 (2) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes